CLINICAL TRIAL: NCT02756312
Title: The Impact of Anesthesia on the Outcome of Supratentorial High- Grade Glioma Patients After Craniotomy
Brief Title: The Impact of Anesthesia on High- Grade Glioma Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Yuming Peng, Professor, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ChiECRCT-20200049
Record Dates: First submitted 2016-04-27; First posted 2016-04-29 (Estimated); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Anesthesia, Outcome, High-grade Glioma
MeSH Terms: conditions — Glioma | interventions — Anesthesia

STUDY DESIGN:
Intervention Model Description: This is a single centre, randomized, parallel group controlled clinical trial in patients with primary HGG. All eligible patients will be 1:1 randomized to the TIVA or INHA group. The object of the trail is to evaluate the effect of propofol or sevoflurane on the prognosis of supratentorial HGG patients after craniotomy.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The anesthesiologist know the grouping .The subjects and the outcome assesor trained for telephone visit were blinded to the grouping
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intravenous anesthesia (Other): Patients will receive total intravenous anesthesia undergoing brain tumor resection.
  Interventions: Other: IV Anesthesia
- Inhalation anesthesia (Other): Patients will receive volatile inhalational anesthesia undergoing brain tumor resection.
  Interventions: Other: IH anesthesia

INTERVENTIONS:
Other: IV Anesthesia — The patients will receive intravenous anesthesia
  Arms: Intravenous anesthesia
Other: IH anesthesia — The patients will receive inhalation anesthesia
  Arms: Inhalation anesthesia

SUMMARY:
Although bench data and retrospective studies have provided a promising picture of the possible influence of anesthetic technique on the risk of tumor progression and patients mortality, current evidence from RCTs is inadequate to show whether the type of anesthetics might influence tumor progression and patient survival.There are many thousands of patients with a cancer diagnosis undergoing surgery every year, and in the context of biological plausibility, it should lead to the urgent undertaking of RCTs to further evaluate the association between the anesthetic management and patient outcome.

DETAILED DESCRIPTION:
Although bench data and retrospective studies have provided a promising picture of the possible influence of anesthetic technique on the risk of tumor progression and patient mortality, current evidence from RCTs is inadequate to show whether the type of anesthetics might influence the outcome of the patients.There are many thousands of patients with a cancer diagnosis undergoing surgery every year, and in the context of biological plausibility, it should lead to the urgent undertaking of RCTs to further evaluate the association between the anesthetic management and patient outcome.

ELIGIBILITY:
Inclusion Criteria:

1)Magnetic radiology imaging diagnosis of supratentorial high-grade glioma; 2) Patients undergoing tumor resection under selective general anesthesia; 3) Age 18-80 years old; 4) Preoperative KPS < 80; 5) With written informed consent by patients or their relatives.

Exclusion Criteria:

1) History of other operations before; 2) Patients with recurrence and metastasis of gliomas or with malignant tumors of other organs; 3) Emergency operation; 4) Critical condition (ASA grade ≥ V before operation, Appendix 1, Severe liver and kidney dysfunction; 5) Patients with mental illness, severe dementia, language disorder, coma, and end-stage disease, etc.; 6) Pregnant or breastfeeding women; 7) Allergic to study drugs;8) Patients who need electrophysiological monitoring during operation. 9) Patients receiving reoperation with different anesthesia methods will be removed and the patients with the same anesthesia method will be continued to observe; 10) Postoperative pathological result is not high-grade glioma.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
overall survival in18 months | Postoperative 18 months
  overall survival in18 months

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Dong J, Wang D, Sun H, Zeng M, Liu X, Yan X, Li R, Li S, Peng Y. Effect of anesthesia on the outcome of high-grade glioma patients undergoing supratentorial resection: study protocol for a pragmatic randomized controlled trial. Trials. 2022 Sep 27;23(1):816. doi: 10.1186/s13063-022-06716-9. PMID 36167574